CLINICAL TRIAL: NCT00899717
Title: Basis for an Etiological Diagnosis and Treatment of the Chronic TMD-pain: RCT Study
Brief Title: Occlusal Adjustment as Treatment for Chronic Orofacial Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Urbano Santana, Prof., University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/017
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Temporomandibular Joint Disorders; Orofacial Pain
Keywords: Temporomandibular Joint Disorders (TMD); Orofacial pain; Limited mouth opening; Craniomandibular dysfunction syndrome; Axiography; Gnatography; Preferred chewing side; Occlusal adjustment; Selective grinding; Handedness; Bruxism; TMD; Costen's Syndrome; Myofascial pain; TMD treatment; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain; Bruxism; Temporomandibular Joint Dysfunction Syndrome; Pain | interventions — Occlusal Adjustment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Procedure: Occlusal adjustment
- B (Placebo Comparator)
  Interventions: Procedure: Placebo occlusal adjustment

INTERVENTIONS:
Procedure: Occlusal adjustment — modification of occlusal surfaces
  Other Names: Selective grinding; Occlusal reshaping; Occlusal equilibration; Occlusal therapy
  Arms: A
Procedure: Placebo occlusal adjustment — Simulated modification of occlusal surfaces
  Arms: B

SUMMARY:
The purpose of this study is to determine whether occlusal adjustment by selective grinding and/or occlusal addition is an effective treatment of chronic temporomandibular joint disorders.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are very common disorders in daily dentistry and oral and maxillofacial practice. The key symptoms are jaw joint pain and limited mouth opening. Other than trauma, the causes remain unknown; consequently, there are no treatments based on specific etiologies. In our experience, patients can usually receive beneficial occlusal adjustments if these are carefully planned and performed in two steps: (1) elimination of premature contacts, which reduces loads in the temporomandibular joints, and (2) individualized remodeling of lateral anterior guidance to facilitate unilateral alternate chewing. The study will use stratified blocking randomization to blindly assign patients to the real or placebo treatment groups in order to evaluate the null hypothesis (H0) that "Occlusal adjustment of sufficient quality has no effect on chronic pain and/or limited mouth opening in TMD patients."

ELIGIBILITY:
Inclusion Criteria:

* People suitable for inclusion in the study are full dentate patients
* Aged between 18 and 65 years
* Patients with chronic TMD pain (and usually with associated limited mouth opening) for whom occlusal adjustment could achieve normal occlusion, both static and functionally equilibrated

Exclusion Criteria:

* Pregnancy
* Trauma
* Previous TMJ surgery
* Patient refusal to consent to participate in the study or significant concerns about the study
* Limited collaboration
* Concurrent active treatment with orthodontics, and active periodontal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José López-Cedrún Cembranos, MD, DDS, PhD, Principal Investigator — Complejo Hospitalario Universitario de La Coruña; Urbano Santana Penín, MD, DDS, PhD, Study Director — Universidad de Santiago de Compostela
Locations (2):
- Spain (2):
  - Complejo Hospitalario Universitario de La Coruña, A Coruña, La Coruña
  - Facultad de Medicina y Odontología, Santiago de Compostela, La Coruña

RESULTS

PARTICIPANT FLOW:
Groups:
- Real Occlusal Adjustment: Occlusal adjustment : modification of occlusal surfaces
- Sham Occlusal Adjustment: Placebo occlusal adjustment : Simulated modification of occlusal surfaces
Period: Overall Study
Arm/Group | Real Occlusal Adjustment | Sham Occlusal Adjustment
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Occlusal Adjustment | Sham Occlusal Adjustment | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.7 (13.7) | 29.73 (8.61) | 32.1 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Spain | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogic Scale for Pain Intensity (0-10)
Description: The primary outcome was self-reported pain intensity on a 0 to 10 cm visual analog scale considering the temporomandibular disorder side, being 0="No pain" and 10="Worst imaginable pain"
Time Frame: Baseline, immediately after therapy, 3 months and 6 months after therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real Occlusal Adjustment | Placebo Occlusal Adjustment
Number analyzed (Participants) | 10 | 11
units on a scale
  Baseline | 6.52 (1.84) [5.75 to 7.56] | 4.8 (1.99) [2.75 to 7]
  Immediately after therapy | .81 (1.56) | 2.05 (2.07)
  3 months after therapy | 2.25 (2.68) | 3.80 (2.94)
  6 months after therapy | .40 (.97) | 4 (2.31)

2. Secondary Outcome: Symptom Checklist-90-Revised (SCL-90-R®)
Description: Scale name: Global Severity Index. Scale graded from 0 to 4. Scores increases as the symptoms severity increases.
Time Frame: Before and 6 months after therapy
Population: Only tests from 15 participants were suitable because of slow or too many positive responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real | Placebo
Number analyzed (Participants) | 8 | 7
units on a scale
  Baseline Global Severity Index | 1.32 (0.91) | 0.58 (0.54)
  6 months after therapy Global Severity Index | 0.75 (0.5) | 0.51 (0.58)

3. Secondary Outcome: Preferred Chewing Side
Description: The change in the habitual chewing side of each participant across the study
Time Frame: Before and 6 months after therapy
Measure: Number; unit: participants
Groups:
- Real Occlusal Adjustment; Placebo Occlusal Adjustment: Number of patients who changed their habitual chewing side
Arm/Group | Real Occlusal Adjustment | Placebo Occlusal Adjustment
Number analyzed (Participants) | 10 | 11
participants
  Baseline | 0 | 0
  6 months after therapy | 8 | 1

4. Secondary Outcome: Maximum Mouth Opening (mm)
Description: Maximum voluntary unassisted mouth opening
Time Frame: 6 months (before and after therapy) including 4 assessment points: pre-treatment, post-treatment, 3- and 6-month follow up
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Real Occlusal Adjustment | Placebo Occlusal Adjustment
Number analyzed (Participants) | 10 | 11
mm
  Baseline | 41.6 (8.26) | 42.36 (10.55)
  Immediately after therapy | 45.50 (7.89) | 45.07 (10.61)
  3 months after therapy | 47.10 (5.26) | 41.27 (11.31)
  6 months after therapy | 49.20 (7.28) | 41.73 (10.34)

5. Secondary Outcome: Condylar Path Angles
Description: Parasagittal plane condylar path angles tracings in relation to the Frankfort line were made following the Gysi extraoral method.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Placebo Occlusal Adjustment: Placebo occlusal adjustment : Simulated modification of occlusal surfaces
Arm/Group | Real Occlusal Adjustment | Placebo Occlusal Adjustment
Number analyzed (Participants) | 10 | 11
degrees
  Right condylar path angle | 52.33 (10.28) | 49 (8.09)
  Left condylar path angle | 49.20 (11.68) | 48.27 (10.21)
  Pain side condylar path angle | 56.75 (12.62) | 51.09 (9.31)
  Non-pain side condylar path angle | 44.78 (6.87) | 46.18 (8.36)

ADVERSE EVENTS:
Arm/Group | Real Occlusal Adjustment | Sham Occlusal Adjustment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No